CLINICAL TRIAL: NCT04854733
Title: Dual Task Performance of Soccer Referees: Cognitive Task or Motor Task
Brief Title: Motor and Cognitive Dual Task Performance in Sports
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 24.04.2019/59
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-04

CONDITIONS: Task Performance
Keywords: Dual-Task Performance; Task- specific Performance; Sports; Agility; Multiple Object Tracking; Referee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Referees: There will be no interventions. Motor and cognitive assessments will be conducted.
- Athletes: There will be no interventions. Motor and cognitive assessments will be conducted.

SUMMARY:
In this study, it is aimed to examine the dual-task performance of soccer referees. For this purpose, it will be investigated whether the motor or cognitive performance of the referees changes when dual-task is assigned and also whether there are differences in dual-task performance between the referees and athletes with similar training program.

DETAILED DESCRIPTION:
In this study, the motor and cognitive dual-task performances of referees will be evaluated. It also will be investigated whether the referees prioritize one of the performances, motor or cognitive, during the dual-task and whether their role in the competition makes a difference compared to athletes. For this purpose, appropriate motor and cognitive tasks were determined by considering the roles of the referees during the competition.

After completing the Demographic Information Form respectively; Edgren Side Step Agility Test as motor performance assessment, Multiple Object Tracking (MOT) as cognitive performance assessment, and finally Dual-Task evaluation using MOT and Edgren Side Step Agility Test will be applied simultaneously. Dual-task costs will be calculated as a percentage of single-task for both motor and cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* To be a soccer referee who trains for a total of 5 hours two days a week, takes part in a maximum of two competitions a week and has been actively affiliated with the National Football Federation for at least 1 year,
* Being an athlete with similar to soccer referees in terms of sociodemographic and physical characteristics and training program,
* Being between aged 18-30 years.

Exclusion Criteria:

* Not attending weekly trainings regularly,
* Having had a surgical operation in the last year,
* Having a history of trauma in the last 6 months,
* Not being able to communicate,
* Having uncorrected visual deficit and hearing problem.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Soccer referees affiliated with the National Football Federation and athletes with similar to soccer referees in terms of sociodemographic and physical characteristics and training program.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Multiple Object Tracking (MOT) | 20 minutes
  Multiple object tracking (MOT) (4 targets), a computer-based cognitive test, is used. Before the test starts, four of the eight black dots on the white screen are randomly determined by flashing. The participant then follows these moving points and marks the correct points after the black dots stop. The selected correct points are noted and saved as P - Proper selection rate in the participant's file.
  After the MOT test is taught, the test is completed in two different speed parameters (240msec, 300msec) in 10sec x 5 repetitions for each speed.
Edgren Side Step Test | 20 minutes
  It is done to test the individual's agility, side speed, and body control. After 15 minutes of warm-up (dynamic stretching and low-pace forward / side running), the Edgren Side Step Test is explained and shown by the researcher.For testing, 5 cones are placed at 1-meter intervals on a 4-meter wide line on a flat non-slip floor. The participant is asked to wait in the middle line with her legs open. During the 10 seconds test, it is asked to step as quickly as possible to the right and left outer cones. It should be ensured that the face is facing forward and that the feet move sideways. After confirming that the test was performed correctly, the best score in the agility test (distance-meter covered in 10 sec) is recorded by applying 3 repetitions.
Dual Task Assessment | 20 minutes
  After performing the single tasks (Multiple Object Tracking (MOT) and Edgren Side Step Test) separately, participants are taken into double task evaluation. While standing in the starting position of the Edgren Side Stepping Test, the MOT test is opened on the screen placed directly opposite the viewing distance (2-meters). After the flashing of the points to be followed at the beginning of the MOT, the MOT and Edgren Side Step Test are started simultaneously with the movement of the points. At the end of 10 seconds, the distance traveled is recorded in meters and the points of the MOT test are followed by the mouse. Dual-Task Assessment is repeated 3 times for each 2 different MOT speeds and scores are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Oğuz, Phd, Study Director — Marmara University Faculty of Health Sciences; Nilufer Keskin Dilbay, MSc, Principal Investigator — Marmara University Faculty of Health Sciences; Hilal B Can, MSc, Principal Investigator — Marmara University Faculty of Health Sciences
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no a plan to make IPD available.